CLINICAL TRIAL: NCT05741658
Title: An Open-Label, Non-randomized, Multi-center Pilot Study to Evaluate the Safety and Efficacy of 4-week, Daily Oral Use of Dapagliflozin 10mg Tablet in Adults With a Fontan Circulation
Brief Title: The Fontan Dapagliflozin Pilot Study
Acronym: FonDap
Status: Enrolling by invitation | Phase: Phase 4 | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: University of California, Los Angeles (Other); Brett Boyer Foundation (Unknown); AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB00254477; ESR-21-21445 (Other: AstraZeneca)
Record Dates: First submitted 2023-02-14; First posted 2023-02-23 (Actual); Last update posted 2025-12-12 (Actual); Status verified 2025-12

CONDITIONS: Heart Failure
Keywords: Fontan; Sodium-glucose Cotransporter-2 (SGLT2) Inhibitors; Heart failure
MeSH Terms: conditions — Heart Failure | interventions — dapagliflozin

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Dapagliflozin (Other): 4-week, Daily Oral Use of Dapagliflozin 10mg Tablet in Adults with Fontan Circulation
  Interventions: Drug: Dapagliflozin 10mg Tab

INTERVENTIONS:
Drug: Dapagliflozin 10mg Tab — Participants will take one Dapagliflozin 10mg tablet once per day for 4 weeks.

SUMMARY:
The goal of this clinical trial is to study if an investigational study drug called Dapagliflozin could prevent heart failure from getting worse in adults with Fontan circulation. The main questions it aims to answer are:

1. Does Dapagliflozin decrease Fontan pressure?
2. Does Dapagliflozin improve exercise capacity and heart failure symptoms?

Participants will have 4 study visits and 2 follow-up phone calls. The total duration of participation in the study will be up to 5 weeks from the time of screening to the completion of the final safety evaluation. Study procedures include the collection of study-related health information and blood samples, physical examination, exercise testing, total body water assessment, blood laboratory testing, health status survey, safety evaluation phone calls, and home blood pressure monitoring.

DETAILED DESCRIPTION:
Background:

The Fontan palliation is subject to progressive physiologic deterioration over time due to chronic elevation in central venous pressures (CVP), compromised cardiac output, and chronic lymphatic congestion and dysfunction. As a result, in adulthood Fontan patients have high rates of hospitalization of ~30% per year and nearly universally succumb to heart failure in the patients' 40s without heart transplant. Currently, there are no medical therapies of proven benefit in prolonging the lifespan of the Fontan palliation or in improving outcomes in Fontan patients.

Rationale:

Given the unusual physiologic stress established by the Fontan palliation, there is reason to believe that sodium-glucose cotransporter-2 (SGLT2) inhibitors might be uniquely beneficial in this small but growing patient population with an orphan disease process. SGLT2 inhibitors may be beneficial for the following reasons. a) Fontan patients are set up for cardiorenal syndrome. The severe end-organ congestion and increased total body water which characterizes Fontan failure are due to compromised cardiac output and chronically and uniquely elevated CVP. SGLT2 inhibitors appear to be uniquely beneficial in this setting based on findings from Dapagliflozin and Prevention of Adverse Outcomes in Heart Failure (DAPA) trial, CANagliflozin cardioVascular Assessment Study (CANVAS) and Empagliflozin Cardiovascular Outcome Event Trial in Type 2 Diabetes Mellitus Patients. Moreover, Griffin and Rao et al recently demonstrated the benefits of empagliflozin on renal sodium handling resulting in decreases in both plasma volume (which would be anticipated to decrease CVP) and total body water (which would be expected to decrease end-organ parenchymal edema and dysfunction). Based on similar mechanisms of action and similarly beneficial effects of dapagliflozin, the investigators anticipate that benefits will be b) Fontan patients who are overweight have a worse prognosis and SGLT2 inhibitors may facilitate modest weight loss. c) Activation of the Renin-Angiotensin-Aldosterone System (RAAS) has been implicated in the progression of Fontan circulatory deterioration, although clinical trials to investigate this hypothesis have not yielded positive results. In case the RAAS hypothesis is true, SGLT2 inhibitors should decrease renin tone by increasing sodium delivery to the macula densa. d) Fontan physiology frequently deteriorates as a result of progressively worsening ventricular systolic and diastolic function. Activation of inflammatory pathways and cardiac myocyte calcium overload have been implicated in this process in non-Fontan related heart failure, and likely play a role as well in Fontan-related heart failure. Putative anti-inflammatory effects and inhibition of the sodium/hydrogen transporter mediated by SGLT2 inhibition may therefore be of benefit in preventing progressive heart failure in Fontan palliated patients.

Study design rationale:

This is a standard study design for a pilot study to investigate the use of an FDA approved drug, dapagliflozin in a new population, namely that of adult patients with a Fontan circulation. The dose and method of administration will be identical to those currently FDA approved. The Fontan circulation was selected as a study condition as it is characterized by a circulatory state that, at baseline, mimics heart failure (elevated central venous pressure, compromised cardiac output). Given this, the investigators believe the efficacy seen in the general heart failure population will be similarly enjoyed in the Fontan population. This study is designed to define more closely the physiologic changes which dapagliflozin create in the Fontan circulation, with the goal of providing data in support of a future larger study of the drug in this population with clinical endpoints.

Study objectives:

The primary objective is to determine the efficacy (as assessed by changes in peripheral venous pressure (PVP) measured by manometry) of Dapagliflozin in decreasing CVPs in Fontan patients. The secondary objective is to Investigate the impact of Dapagliflozin on CVP, total body water, exercise capacity, and patient-reported health status in Fontan patients.

Sample size:

Based on variability in PVP in Fontan patients as published by Tan et al(14) 18.4 + 5 millimeters of mercury (mmHg) with a drop of 4 mmHg is assumed to be of clinical significance, with alpha = 5% powered at 80% a total of 26 patients would be required. Allowing for ~10%, this yields a target recruitment of 29 patients.

Statistical analyses:

For the primary endpoint, the investigators will compare the change in PVP and total body water at baseline and at the end of the study period for differences using ANOVA for the primary endpoint. For the secondary endpoint, the investigators will compare change in total body water, maximum rate of oxygen your body is able to use during exercise, the minute ventilation/carbon dioxide production, oxygen pulse, and oxygen uptake efficiency slope assessed during cardiopulmonary exercise testing, patient reported health status outcome metric score as assessed by Adult Congenital Heart Disease Patient Reported Outcome (ACHD PRO) between baseline and at the end of the study period using ANOVA for the secondary endpoints.

ELIGIBILITY:
Inclusion Criteria:

For inclusion in the study subjects should fulfil the following criteria based on local regulations:

1. Provision of informed consent prior to any study specific procedures
2. Female and/or male subjects aged ≥18 years
3. Subjects with Fontan circulation (in the opinion of the PI)
4. Subjects with clinical stability for 6 months preceding enrollment (in the opinion of the PI)
5. Subjects with no planned changes in medical therapy in the 1 months after enrollment
6. Subjects with no planned interventional procedures in the 1 months after enrollment
7. Negative pregnancy test (urine or serum) for female subjects of childbearing potential.
8. Female subjects must be 1 year post-menopausal, surgically sterile, or using an acceptable method of contraception (an acceptable method of contraception is defined as a barrier method in conjunction with a spermicide) for the duration of the study (from the time the subjects sign consent) and for 3 months after the last dose of Drug A/matching placebo to prevent pregnancy. In addition, oral contraceptives, approved contraceptive implant, long-term injectable contraception, intrauterine device, or tubal ligation are allowed. Oral contraception alone is not acceptable; additional barrier methods in conjunction with spermicide must be used.
9. Male subjects must be surgically sterile or using an acceptable method of contraception (defined as barrier methods in conjunction with spermicides) for the duration of the study (from the time the subjects sign consent) and for 3 months after the last dose of Drug A/matching placebo to prevent pregnancy in a partner.
10. Subjects who are blood donors should not donate blood during the study and for 3 months following the subject's last dose of dapagliflozin.

Exclusion Criteria:

Subjects should not enter the study if any of the following exclusion criteria are fulfilled:

1. Involvement in the planning and/or conduct of the study (applies to both Investigator staff and/or staff at the study site)
2. Previous enrollment or randomisation in the present study
3. Participation in another clinical study with an investigational product during the last 6 months
4. Pregnancy or breast feeding or desire to become pregnant or breast feed during the study period
5. Hospitalization within 6 months prior to enrollment
6. Arrhythmia requiring change in therapy within 6 months prior to enrollment
7. Interventional procedure of any kind (including cardioversion) within 6 months prior to enrollment
8. Difficulty with upper extremity IV placement in the past
9. Known obstruction anywhere within the venous circulation including at the level of the Glenn or Fontan anastomosis or within the pulmonary vasculature.
10. Symptomatic hypotension or systemic systolic blood pressure of <95 millimeters of mercury (mmHg)
11. Estimated glomerular filtration rate of <25ml per minute per 1.73m2 body surface area as assessed by Modification of Diet in Renal Disease (MDRD) calculation
12. Prior use of SGLT2 inhibitors with intolerable side effects
13. Type 1 diabetes
14. Inability to comply with the study protocol
15. Lack of English-proficiency
16. History of hypersensitivity to SGLT2 inhibitors
17. Severe hepatic impairment defined as a Model for End-stage Liver Disease (MELD) XI score of >10

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Estimated)
Dates: Start 2023-11-08 (Actual); Primary Completion 2026-02 (Estimated); Study Completion 2026-02 (Estimated)

PRIMARY OUTCOMES:
Peripheral venous pressure (millimeters of mercury) at rest measured by manometry | From baseline at week 0 and to follow up at week 4
  To investigate the impact of Dapagliflozin on changing central venous pressure in Fontan patients

SECONDARY OUTCOMES:
Total body water (liter) as measured by bioelectrical impedance analyzer | From baseline at week 0 and to follow up at week 4
  To Investigate the impact of Dapagliflozin on changing total body water
Maximal oxygen uptake (milliliters/kilograms/minutes) as measured by cardiopulmonary exercise test | From baseline at week 0 and to follow up at week 4
  To Investigate the impact of Dapagliflozin on maximal oxygen uptake
oxygen pulse (milliliters oxygen per beat per kilogram) as measured by cardiopulmonary exercise test | From baseline at week 0 and to follow up at week 4
  To Investigate the impact of Dapagliflozin on oxygen pulse
ventilator efficiency slope (no unit) as measured by cardiopulmonary exercise test | From baseline at week 0 and to follow up at week 4
  To Investigate the impact of Dapagliflozin on ventilator efficiency slope
oxygen uptake efficiency slope (no unit) as measured by cardiopulmonary exercise test | From baseline at week 0 and to follow up at week 4
  To Investigate the impact of Dapagliflozin on oxygen uptake efficiency slope
Peripheral venous pressure (mmHg) at exercise measured by manometry | From baseline at week 0 and to follow up at week 4
  To investigate the impact of Dapagliflozin on changing central venous pressure in Fontan patients
Patient reported health status as measure by the ACHD PRO metric score | From baseline at week 0 and to follow up at week 4
  To Investigate the impact of Dapagliflozin on patient-reported health status in Fontan patients The overall score ranges from 0 to 100, with 0 being worst and 100 being excellent.

CONTACTS AND LOCATIONS:
Overall Officials: Ari Cedars, Principal Investigator — Johns Hopkins University
Locations (1):
- Ronald Reagan UCLA Medical Center, Los Angeles, California, United States

REFERENCES:
- [Background] Akintoye E, Miranda WR, Veldtman GR, Connolly HM, Egbe AC. National trends in Fontan operation and in-hospital outcomes in the USA. Heart. 2019 May;105(9):708-714. doi: 10.1136/heartjnl-2018-313680. Epub 2018 Oct 30. PMID 30377261
- [Background] Rychik J, Atz AM, Celermajer DS, Deal BJ, Gatzoulis MA, Gewillig MH, Hsia TY, Hsu DT, Kovacs AH, McCrindle BW, Newburger JW, Pike NA, Rodefeld M, Rosenthal DN, Schumacher KR, Marino BS, Stout K, Veldtman G, Younoszai AK, d'Udekem Y; American Heart Association Council on Cardiovascular Disease in the Young and Council on Cardiovascular and Stroke Nursing. Evaluation and Management of the Child and Adult With Fontan Circulation: A Scientific Statement From the American Heart Association. Circulation. 2019 Aug 6;140(6):e234-e284. doi: 10.1161/CIR.0000000000000696. Epub 2019 Jul 1. PMID 31256636
- [Background] Rychik J. Forty years of the Fontan operation: a failed strategy. Semin Thorac Cardiovasc Surg Pediatr Card Surg Annu. 2010;13(1):96-100. doi: 10.1053/j.pcsu.2010.02.006. No abstract available. PMID 20307870
- [Background] McMurray JJV, Solomon SD, Inzucchi SE, Kober L, Kosiborod MN, Martinez FA, Ponikowski P, Sabatine MS, Anand IS, Belohlavek J, Bohm M, Chiang CE, Chopra VK, de Boer RA, Desai AS, Diez M, Drozdz J, Dukat A, Ge J, Howlett JG, Katova T, Kitakaze M, Ljungman CEA, Merkely B, Nicolau JC, O'Meara E, Petrie MC, Vinh PN, Schou M, Tereshchenko S, Verma S, Held C, DeMets DL, Docherty KF, Jhund PS, Bengtsson O, Sjostrand M, Langkilde AM; DAPA-HF Trial Committees and Investigators. Dapagliflozin in Patients with Heart Failure and Reduced Ejection Fraction. N Engl J Med. 2019 Nov 21;381(21):1995-2008. doi: 10.1056/NEJMoa1911303. Epub 2019 Sep 19. PMID 31535829
- [Background] Zinman B, Wanner C, Lachin JM, Fitchett D, Bluhmki E, Hantel S, Mattheus M, Devins T, Johansen OE, Woerle HJ, Broedl UC, Inzucchi SE; EMPA-REG OUTCOME Investigators. Empagliflozin, Cardiovascular Outcomes, and Mortality in Type 2 Diabetes. N Engl J Med. 2015 Nov 26;373(22):2117-28. doi: 10.1056/NEJMoa1504720. Epub 2015 Sep 17. PMID 26378978
- [Background] Radholm K, Figtree G, Perkovic V, Solomon SD, Mahaffey KW, de Zeeuw D, Fulcher G, Barrett TD, Shaw W, Desai M, Matthews DR, Neal B. Canagliflozin and Heart Failure in Type 2 Diabetes Mellitus: Results From the CANVAS Program. Circulation. 2018 Jul 31;138(5):458-468. doi: 10.1161/CIRCULATIONAHA.118.034222. PMID 29526832
- [Background] Figtree GA, Radholm K, Barrett TD, Perkovic V, Mahaffey KW, de Zeeuw D, Fulcher G, Matthews DR, Shaw W, Neal B. Effects of Canagliflozin on Heart Failure Outcomes Associated With Preserved and Reduced Ejection Fraction in Type 2 Diabetes Mellitus. Circulation. 2019 May 28;139(22):2591-2593. doi: 10.1161/CIRCULATIONAHA.119.040057. Epub 2019 Mar 17. No abstract available. PMID 30882240
- [Background] Griffin M, Rao VS, Ivey-Miranda J, Fleming J, Mahoney D, Maulion C, Suda N, Siwakoti K, Ahmad T, Jacoby D, Riello R, Bellumkonda L, Cox Z, Collins S, Jeon S, Turner JM, Wilson FP, Butler J, Inzucchi SE, Testani JM. Empagliflozin in Heart Failure: Diuretic and Cardiorenal Effects. Circulation. 2020 Sep 15;142(11):1028-1039. doi: 10.1161/CIRCULATIONAHA.120.045691. Epub 2020 May 15. PMID 32410463
- [Background] Neal B, Perkovic V, Mahaffey KW, de Zeeuw D, Fulcher G, Erondu N, Shaw W, Law G, Desai M, Matthews DR; CANVAS Program Collaborative Group. Canagliflozin and Cardiovascular and Renal Events in Type 2 Diabetes. N Engl J Med. 2017 Aug 17;377(7):644-657. doi: 10.1056/NEJMoa1611925. Epub 2017 Jun 12. PMID 28605608
- [Background] Packer M, Anker SD, Butler J, Filippatos G, Zannad F. Effects of Sodium-Glucose Cotransporter 2 Inhibitors for the Treatment of Patients With Heart Failure: Proposal of a Novel Mechanism of Action. JAMA Cardiol. 2017 Sep 1;2(9):1025-1029. doi: 10.1001/jamacardio.2017.2275. PMID 28768320
- [Background] Koyani CN, Plastira I, Sourij H, Hallstrom S, Schmidt A, Rainer PP, Bugger H, Frank S, Malle E, von Lewinski D. Empagliflozin protects heart from inflammation and energy depletion via AMPK activation. Pharmacol Res. 2020 Aug;158:104870. doi: 10.1016/j.phrs.2020.104870. Epub 2020 May 17. PMID 32434052
- [Background] Packer M. Interplay of adenosine monophosphate-activated protein kinase/sirtuin-1 activation and sodium influx inhibition mediates the renal benefits of sodium-glucose co-transporter-2 inhibitors in type 2 diabetes: A novel conceptual framework. Diabetes Obes Metab. 2020 May;22(5):734-742. doi: 10.1111/dom.13961. Epub 2020 Feb 20. PMID 31916329
- [Background] Cedars AM, Ko JM, John AS, Vittengl J, Stefanescu-Schmidt AC, Jarrett RB, Kutty S, Spertus JA. Development of a Novel Adult Congenital Heart Disease-Specific Patient-Reported Outcome Metric. J Am Heart Assoc. 2020 Jun 2;9(11):e015730. doi: 10.1161/JAHA.119.015730. Epub 2020 May 16. PMID 32419592
- [Background] Tan W, Small A, Gallotti R, Moore J, Aboulhosn J. Peripheral venous pressure accurately predicts central venous pressure in the adult Fontan circulation. Int J Cardiol. 2021 Mar 1;326:77-80. doi: 10.1016/j.ijcard.2020.11.007. Epub 2020 Nov 13. PMID 33189798
- [Background] Kushner RF, Schoeller DA. Estimation of total body water by bioelectrical impedance analysis. Am J Clin Nutr. 1986 Sep;44(3):417-24. doi: 10.1093/ajcn/44.3.417. PMID 3529918
- [Background] Bedogni G, Malavolti M, Severi S, Poli M, Mussi C, Fantuzzi AL, Battistini N. Accuracy of an eight-point tactile-electrode impedance method in the assessment of total body water. Eur J Clin Nutr. 2002 Nov;56(11):1143-8. doi: 10.1038/sj.ejcn.1601466. PMID 12428182